CLINICAL TRIAL: NCT04212728
Title: Treatment of Knee Osteoarthritis With Autologous Adipose-derived Mesenchymal Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Principal Investigator, Peiwen Lian, Peiwen Lian Ph.D, Yantai Yuhuangding Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-003
Record Dates: First submitted 2019-12-26; First posted 2019-12-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMSCs plus PRP group (Experimental): Three intra-articular injections in total and autologous adipose-derived mesenchymal stem cells (AMSCs) suspended in 3 ml autologous platelet rich plasma (PRP) for each injection. Time-points for intervention: 1) initial injection; 2) 3 months following initial injection; 3) 6 months following initial injection.
  Interventions: Biological: Auotologous AMSCs plus autologous PRP
- PRP group (Active Comparator): Three intra-articular injections in total and 3 ml autologous platelet rich plasma (PRP) for each injection. Time-points for intervention: 1) initial injection; 2) 3 months following initial injection; 3) 6 months following initial injection.
  Interventions: Biological: Auotologous PRP

INTERVENTIONS:
Biological: Auotologous AMSCs plus autologous PRP — 150 mL subcutaneous abdominal adipose tissue will be harvested via liposuction . AMSCs will be isolated and cultured from adipose tissue. Before injection, 30 mL of blood will be collected from each patient to produce 3ml PRP by cenrifugation.Cultured AMSCs will be collected and suspended by 3ml autologous PRP.
  Arms: AMSCs plus PRP group
Biological: Auotologous PRP — 30 mL of blood will be collected from each patient to produce 3ml PRP by cenrifugation.
  Arms: PRP group

SUMMARY:
The purpose of this study is to explore the efficacy and safety of autologous adipose-derived mesenchymal stem cells (AMSCs) plus autologous platelet rich plasma (PRP) in the treatment of severe knee osteoarthritis.

DETAILED DESCRIPTION:
This is a single centered, randomized, single blind phase II clinical study. Patients will be divided into two groups of case and control. Patients of case group will receive intra-articular injection of autologous AMSCs suspended in 3 ml autologous PRP for 3 times, patients of control group will receive intra-articular injection of 3 ml of autologous PRP for 3 times. The investigators designed this clinical study to evaluate therapeutic effects of AMSCs in patients with severe knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Kellgren and Lawrence grade II-IV primary osteoarthritis as determined by X-ray.
2. Subject's pain score is 8-13 points (Lequesne's index).
3. Ages between 40-70 years.
4. Signed informed consent from the subject.

Exclusion Criteria:

1. Subject infected with hepatitis B, hepatitis C, HIV, syphilis or HTLV
2. Subject not suitable for liposuction surgery.
3. Subject with hypersensitivity/allergy to anesthetic.
4. Subject's creatinine values higher than 1.6mg/dl.
5. Subject with body mass index, BMI over 30.
6. Subject's studied knee treated with intra-articular injection therapy within 6 months prior to screen.
7. Subject has undergone surgery on studied knee, including fracture surgery, arthroscopic surgery, meniscus repair surgery, or cruciate ligament reconstruction surgery.
8. Subject enrolled in any other cell therapy studies within the past 30 days.
9. Subject who the investigator considers inappropriate for the clinical trial due to any other reasons than those listed above.
10. Subject has a history of gouty arthritis, septic arthritis, rheumatoid arthritis and any other autoimmune arthritis of the knee joint.
11. Subject has had major medical problems in vital organs, such as; heart, liver, kidney, or lung.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Physical function change | From before randomization until 3, 6, and 12 months after treatment start.
  Evaluation the physical function change measured by the Western Ontario and McMaster Universities Arthritis Index (WOMAC). The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations.
Change in pain density | From before randomization until 3, 6, and 12 months after treatment start.
  Evaluation the changing of pain density measured by Visual Analogue Scale. Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.

SECONDARY OUTCOMES:
Cartilage repair | From before randomization until 3, 6, and 12 months after treatment start.
  Evaluation of cartilage repair under MRI. Recht criterion was used for grading articular cartilage injury of knee joint, including 0-IV grade, in which: 0 grade, normal articular cartilage, no obvious abnormal signal was found; 1 grade, the layered structure of cartilage disappeared, and there were focal low signal areas, but the surface was smooth; 2 grade, the surface of cartilage was irregular, the depth of cartilage injury was less than 50% cartilage thickness; 3 grade, the surface of cartilage was heavy. The degree of injury is irregular, the depth of injury is more than 50% of the thickness of cartilage or through the whole layer, but the surface of cartilage is not completely exfoliated; Grade IV, full-thickness cartilage defect, articular cartilage injury deep to the cortex, subchondral bone exposed.
Change in MOS item short from health survey(SF-36) | From before randomization until 3, 6, and 12 months after treatment start.
  Evaluation of the health-related quality of life change Measured by MOS item short from health survey(SF-36) after each cell injection. SF-36 is a self-administered questionnaire comprising 36-items measuring eight dimensions of general HRQOL: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items).These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.
Change in Lequesne Index | From before randomization until 3, 6, and 12 months after treatment start.
  Evaluation of severity of knee symptoms Lequesne Index includes the measurement of pain (5 items), walking distance (2 items), and activities of daily living (4 items). Maximal score is 24 and higher scores represent worse function
Change in knee society score (KSS) | From before randomization until 3, 6, and 12 months after treatment start.
  The knee society score is divided into four parts: it consists of the ''Symptoms''(25 points), the ''Patient satisfaction''(40 points), the ''Patient expectation''(15 points) and the ''Functional activities''(100 points). Each part will be evaluated separately.Higher scores indicate better knee score/satisfaction/functioning or higher expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Peiwen Lian, PhD, Study Director — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China